CLINICAL TRIAL: NCT06079983
Title: A Phase 3, Multicenter, Randomized, Open-Label, Active-Controlled Trial Of JSKN003 Versus Treatment Of Physician'S Choice For HER2-low, Unresectable and/or Metastatic Breast Cancer Subjects
Brief Title: JSKN003 Versus Treatment Of Physician'S Choice For HER2-low, Unresectable and/or Metastatic Breast Cancer Subjects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-302
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Gemcitabine; Injections; Vinorelbine; Paclitaxel; Docetaxel; eribulin

STUDY DESIGN:
Intervention Model Description: A Phase 3, Multicenter, Randomized, Open-Label, Active-Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JSKN003 (Experimental): Administered intravenously according to protocol.
  Interventions: Drug: JSKN003
- The chemotherapy chosen by the investigator (Active Comparator): The mono-chemotherapy drugs selected by the investigators included capecitabine, gemcitabine, vinorelbine, docetaxel, albumin-bound paclitaxel, or eribulin. The option should be determined before randomization.
  Interventions: Drug: Capecitabine tablets; Drug: Gemcitabine hydrochloride for injection; Drug: Vinorelbine tartrate injection; Drug: Paclitaxel for injection (albumin-bound type); Drug: Docetaxel injection; Drug: Eribulin mesylate injection

INTERVENTIONS:
Drug: JSKN003 — Administered intravenously according to protocol.
  Arms: JSKN003
Drug: Capecitabine tablets — Administered according to protocol, as one option for investigator's choice (determined before randomization).
  Arms: The chemotherapy chosen by the investigator
Drug: Gemcitabine hydrochloride for injection — Administered according to protocol, as one option for investigator's choice (determined before randomization).
  Arms: The chemotherapy chosen by the investigator
Drug: Vinorelbine tartrate injection — Administered according to protocol, as one option for investigator's choice (determined before randomization).
  Arms: The chemotherapy chosen by the investigator
Drug: Paclitaxel for injection (albumin-bound type) — Administered according to protocol, as one option for investigator's choice (determined before randomization).
  Arms: The chemotherapy chosen by the investigator
Drug: Docetaxel injection — Administered according to protocol, as one option for investigator's choice (determined before randomization).
  Arms: The chemotherapy chosen by the investigator
Drug: Eribulin mesylate injection — Administered according to protocol, as one option for investigator's choice (determined before randomization).
  Arms: The chemotherapy chosen by the investigator

SUMMARY:
This study is a randomized controlled, open-label, multicenter phase III clinical study evaluating the efficacy and safety of chemotherapy selected by investigator JSKN003 s in subjects with recurrent or metastatic breast cancer who have previously failed first- or second-line chemotherapy in subjects with recurrent or metastatic breast cancer who have failed prior first- or second-line chemotherapy.

The study planned to enroll 408 subjects in a 1:1 ratio and stratified block randomization method assigned to:

* Experimental group: JSKN003 monotherapy
* Control group: investigator's chosen chemotherapy drug (capecitabine, gemcitabine, vinorelbine, docetaxel, albumin-bound paclitaxel, or eribulin) monotherapy

DETAILED DESCRIPTION:
This study is a randomized controlled, open-label, multicenter phase III clinical study evaluating the efficacy and safety of chemotherapy selected by investigator JSKN003 s in subjects with recurrent or metastatic breast cancer who have previously failed first- or second-line chemotherapy in subjects with recurrent or metastatic breast cancer who have failed prior first- or second-line chemotherapy.

The study planned to enroll 408 subjects in a 1:1 ratio and stratified block randomization method assigned to:

* Experimental group: JSKN003 monotherapy
* Control group: investigator's chosen chemotherapy drug (capecitabine, gemcitabine, vinorelbine, docetaxel, albumin-bound paclitaxel, or eribulin) monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject is able to understand the informed consent form, voluntarily participate and sign the informed consent form.

  2. The subject ≥ 18 years old on the day of signing the informed consent form, male or female.

  3. Unresectable locally recurrent or metastatic breast cancer, previous histopathological reports of HER2 IHC 1+ or 2+ and ISH-, previous histopathological reports have not been diagnosed as HER2 IHC 3+ or 2+ and ISH+.

  4. Have received at least 1 to 2 lines of chemotherapy regimens for breast cancer in the relapse/metastatic stage.

  5. Willing to provide sufficient archived tumor pathology specimens for central laboratory detection of HER2 status.

  6. Documented radiographic disease progression (during or after the most recent treatment).

  7. At least one extracranial measurable lesion at baseline according to RECIST 1.1 criteria.

  8. Expected survival ≥ 3 months. 9. ECOG score of 0 or 1 within 14 days prior to administration. 10. Female subjects of childbearing potential or male subjects of fertile partner consent to use highly effective contraception from the signing of informed consent.

  11. Laboratory tests within 14 days before administration and cardiac function tests within 28 days meet the criteria.

  12. Have sufficient elution of previous treatment before administration.

Exclusion Criteria:

* 1. Untreated, or unstable brain parenchymal metastases, spinal cord metastases or compression, cancerous meningitis.

  2. Patients with only skin lesions as target lesions. 3. Those with a history of other primary malignant tumors within 5 years before administration.

  4. Selection of the control drug by the investigator who is not suitable for the protocol prescribed.

  5. Previous use of antibody conjugates containing topoisomerase I inhibitors. 6. There is a third gap fluid that cannot be controlled by drainage, etc. 7. Previous or current interstitial pneumonia/lung disease requiring systemic hormone therapy.

  8. Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors that affect oral administration and absorption of the drug.

  9. Previous or current autoimmune disease. 10. Have uncontrolled comorbidities. 11. The toxicity of previous antitumor therapy has not been restored to grade ≤1 (NCI-CTCAE v5.0).

  12. History of previous immunodeficiency. 13. History of life-threatening allergic reactions or known ≥ grade 3 allergy to any component or excipient in the investigational pharmaceutical formulation.

  14. Other conditions that the investigators believe will affect the safety or adherence to drug treatment in this study, including but not limited to psychiatric disorders, alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to approximately 3 years after the first enrollment
  PFS evaluated by BICR according to RECIST v1.1 criteria is defined as the time from randomization to the first recorded disease progression or death from any cause as a result of BICR evaluation according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival（OS） | up to approximately 3 years after the first enrollment
  OS, defined as the time from randomization to death from any cause;
Objective Response Rate (ORR) | up to approximately 3 years after the first enrollment
  BICR and investigators were judged according to RECIST v1.1 criteria ，objective response rate (ORR), defined as the proportion of participants achieving a complete response (CR) or partial response (PR) according to RECIST v1.1 criteria;
Duration of Response (DOR) | up to approximately 3 years after the first enrollment
  BICR and investigators were judged according to RECIST v1.1 criteria，Duration of response (DoR), defined as the time from the first recorded response (CR/PR) to the first documented disease progression (PD) or death from any cause;

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Jiong Wu, Principal Investigator — Fudan University
Locations (87):
- China (87):
  - Erwei Song, Guangzhou, Guangdong
  - Jiong Wu, Shanghai, Shanghai Municipality
  - Anyang Cancer Hospital, Anyang
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Luhe Hospital, Beijing
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University Cancer Hospital, Beijing
  - The First Affiliated Hospital of China Medical University, Beijing
  - The First Medical Center of the General Hospital of the People's Liberation Army Chinese People's Liberation Army, Beijing
  - Bethune First Hospital of Jilin University, Changchun
  - Jilin Provincial Cancer Hospital, Changchun
  - The First People's Hospital of Changde, Changde
  - Central South University Xiangya Hospital, Changsha
  - Hunan Cancer Hospital, Changsha
  - Affiliated Hospital of Chengde Medical University, Chengde
  - Sichuan Cancer Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Cancer Hospital of Chongqing University, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Provincial Hospital, Fuzhou
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The Affiliated Hospital of Guangdong Medical University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guanzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Run Run Shaw Hospital affiliated to Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou
  - Zhejiang Cancer Hospital, Hanzhou
  - Harbin Medical University Cancer Hospital, Ha’erbin
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of University of South China, Hengyang
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jiangmen Central Hospital, Jiangmen
  - Shandong Cancer Hospital, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Yunnan Cancer Hospital, Kunming
  - Gansu Provincial Cancer Hospital, Lanzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - Linyi Cancer Hospital, Linyi
  - Linyi People's Hospital, Linyi
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Meizhou People's Hospital, Meizhou
  - Jiangxi Provincial Cancer Hospital, Nanchang
  - The Third Hospital of Nanchang, Nanchang
  - Jiangsu Provincial Cancer Hospital, Nanjing
  - Jiangsu Provincial People's Hospital, Nanjing
  - Cancer Hospital Affiliated to Guangxi Medical University, Nanning
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning
  - The Second People's Hospital of Neijiang, Neijiang
  - Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Cancer Hospital, Shanghai
  - Cancer Hospital Affiliated to Shantou University School of Medicine, Shantou
  - The People's Hospital of Northern Guangdong, Shaoguan
  - Liaoning Cancer Hospital, Shengyang
  - Suining Central Hospital, Suining
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Bethune Hospital, Taiyuan
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Zhejiang Taizhou Hospital, Taizhou
  - Tianjin Cancer Hospital, Tianjin
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi
  - Hubei Provincial Cancer Hospital, Wuhan
  - People's Hospital of Wuhan University, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - Affiliated Hospital of Qinghai University, Xining
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Yongzhou Central Hospital in Hunan Province, Yongzhou
  - The First People's Hospital of Zhaoqing, Zhaoqing
  - Henan Provincial Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: No